CLINICAL TRIAL: NCT06781398
Title: Robotic Surgery in the Treatment of Deep Endometriosis: Da Vinci Vs HUGO RAS Compared
Brief Title: Robotic Surgery in the Treatment of Deep Endometriosis: Da Vinci Vs HUGO RAS Comparison
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ROBOTENDO
Record Dates: First submitted 2024-12-03; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-10

CONDITIONS: Deep Endometriosis
Keywords: endometriosis; gynaecology; surgery; Da Vinci; HUGO RAS
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim is to clarify whether both surgical approaches represent, equivalently, a good treatment for the management of patients with deep endometriosis who are candidates for surgery, or whether there are any differences between the two methods, and, if so, how they differ

DETAILED DESCRIPTION:
Numerous studies have shown how surgical excision of deep endometriosis nodules improves pain and quality of life. Robotic-assisted laparoscopic surgery has been employed for the treatment of deep endometriosis. While the Da Vinci System is widely used for the surgical treatment of endometriosis, with good results, the available data regarding the benefits of the HUGO RAS System, however, are limited, given the recent introduction of this method in gynecology, and particularly in the treatment of endometriosis. The aim of the study is to investigate whether the robotic surgical approach using HUGO RAS is noninferior to that performed using Da Vinci in terms of operative time (docking + surgical time) in the surgical treatment of patients with endometriosis

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55 years;
* Pelvic ultrasound and/or radiologic (MRI/CT scan with rectal insufflation) diagnosis of endometriosis
* Indication for surgery (symptomatic despite or refractory to medical therapy, and/or with critical bowel stenosis or urinary stenosis, and/or infertile awaiting medically assisted procreation (PMA) treatment or with previous failed assisted fertilization attempts);
* ASA (American Society of Anesthesiologists physical status classification) class between 1 and 3;
* Acquisition of consent to undergo surgical treatment;
* Acquisition of consent for study participation and data processing

Exclusion Criteria:

- Past or current diagnosis of gynecologic oncologic pathology.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who are candidates for surgery with minimally invasive approach for endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
The robotic surgical approach using HUGO RAS is noninferior to that performed using Da Vinci in terms of operative time (docking + surgical time) in the surgical treatment of patients with endometriosis | During surgery
  Compare the two surgical techniques by evaluating the operative time (expressed in minutes), which includes docking and surgical time.
  Docking is defined as the time required to move the robotic arms into the operative field, place them in their respective port sites, and insert the robotic instruments into the abdomen.
  Surgical time is from the end of docking to suturing the laparoscopic/laparotomy breaches.

SECONDARY OUTCOMES:
Conversion rate to laparoscopy or laparotomy | During surgery
  Conversion to laparoscopy or laparotomy, based on intraoperative assessment of the clinical picture
Intra-operative and post-operative complication rates; need for complication treatment | Perioperative and at 3 months
  Intraoperative complications (incidental injury to organs and structures, incoercible bleeding) classified by ClassIntra System (iAE); postoperative complications (anemia, postoperative fever, hemoperitoneum, bowel perforation), according to Clavien-Dindo classification; treatment of complications (GRC transfusion, reintervention, interventional procedures)
Ergonomics for the surgeon | During surgery
  Ergonomics of the two robotic approaches established through the Rapid Upper Limb Assessment (RULA) system that allows through the compilation of a score, rapid assessment of the load on the neck and upper limb. The risk of work-related disorders is calculated in a score from 1 (low) to 7 (high)
Entity of postoperative pain | Perioperative and at 3 and 12 months
  Postoperative pain assessed as maximum value recorded by numeric rating scale (NRS), from 0 to 10, corresponding to 'no pain' and 'worst pain imaginable' respectively
Hospitalization time | From the day of admission to the day of discharge, an average of 1 year
  Hospitalization time
Assessment of pain and quality of life | At 3 and 12 months after surgery
  Pain assessment and change in quality of life, assessed by administration of NRS scale, from 0 to 10, corresponding to 'no pain' and 'worst pain imaginable' respectively
Assessment of pain and quality of life | At 3 and 12 months after surgery
  Pain assessment and change in quality of life, assessed by administration of quality of life questionnaire (EHP-30, Endometriosis-related health profile), scored from 0 to 100, with 0 being the best outcome and 100 the worst outcome
Symptomatological and/or anatomical recurrence | At 12 months after surgery
  Clinical or anatomical resumption of disease by gynecological examination, recent pathological history, pelvic ultrasound, and possible radiological methods such as nuclear magnetic resonance imaging (NMR)

CONTACTS AND LOCATIONS:
Overall Officials: Diego Raimondo, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (2):
- Italy (2):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Università Cattolica del Sacro Cuore, Roma, Roma